CLINICAL TRIAL: NCT07084584
Title: A Phase 1/2, Open-label, Dose-Escalation and Dose-Expansion Cohort Study of GB3226 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: An Open-label, Dose-Escalation and Dose-Expansion Study of GB3226 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GB3226-DEV-001
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): Cohort A: Patients must not be receiving any weak, moderate, or strong CYP3A4 inhibitors/inducers. Patients who were receiving a CYP3A4 inhibitor/inducer must have discontinued the medication at least 7 days prior to enrolment
  Interventions: Drug: GB3226
- Cohort B (Experimental): Cohort B: Patients must be receiving a strong CYP3A4 inhibitor for antifungal prophylaxis (e.g. parconazole, itraconazole, ketoconazole, or voriconazole) for at least 7 days prior to enrolment and while on GB3226 treatment. Patients must not be receiving any other strong CYP3A4 inhibitors/inducers.
  Interventions: Drug: GB3226
- Cohort C (Experimental): Cohort C: Patients must be receiving a moderate CYP3A4 inhibitor for antifungal prophylaxis (e.g., isavuconazole, fluconazole) for at least 7 days prior to enrolment and while on GB3226. Patients must not be receiving any other strong or moderate CYP3A4 inhibitors/inducers.
  Interventions: Drug: GB3226

INTERVENTIONS:
Drug: GB3226 — GB3226: Dual inhibitor of ENL-YEATS and FLT3 pathways Administration: Oral, daily dosing in 28-day cycles

SUMMARY:
Study GB3226-DEV-001 is a Phase 1/2, open-label, dose-escalation and expansion study of GB3226 in the treatment of relapsed or refractory acute myeloid leukaemia

DETAILED DESCRIPTION:
Study GB3226-DEV-001 is a Phase 1/2, open-label, dose-escalation and expansion study of GB3226 in the treatment of relapsed or refractory acute myeloid leukemia. Adult patients aged ≥18 years of age are planned to be enrolled. GB3226 will be administered once daily orally (PO) in 28-day cycles, with the first study drug dose administered on Cycle 1 Day 1 (C1D1). Up to a total of three separate patient cohorts will be explored (GB3226 without a CYP3A4 inhibitor, GB3226 with a strong CYP3A4 inhibitor and, if indicated, a cohort of GB3226 with a moderate CYP3A4 inhibitor).

ELIGIBILITY:
Eligible participants are males and female aged 18 years or older at screening with relapsed or refractory acute myeloid leukemia Diagnosis

1. Patients in Phase 1 must have active acute myeloid leukemia (bone marrow blasts ≥5% or reappearance of blasts in peripheral blood) as defined by the National Comprehensive Cancer Network (NCCN) in the NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines, Version 3.2024).
2. Phase 2 patients must have documented active acute leukemia (bone marrow blasts ≥5% or reappearance of blasts in peripheral blood) as defined by the NCCN Guidelines for Acute Myeloid Leukemia (Version 3.2024) and may have specific genetic profiles.

   For Phase 2, if inclusion is restricted to specific genetic subtypes, mutational status will be assessed locally for initial eligibility determination and confirmed by central laboratory testing. Patients with mutational status not confirmed centrally, or with final pathology or flow cytometry reports indicating <5% bone marrow blasts, will be replaced to ensure adequate enrolment for the primary efficacy analyses.

   Disease Status
3. Recurrent or refractory AML, as defined by standardized criteria (for example, European LeukemiaNet criteria (Döhner 2022); International Working Group criteria (Cheson 2003)) after standard of care therapy, including but not limited to one or two cycles of intensive chemotherapy, or venetoclax combinations. Patients with persistent leukemia after initial therapy or with recurrence of leukemia at any time after achieving a response during or after the course of treatment (including allogeneic HSCT) are eligible. Refractory or relapsed leukemia is defined by presence of ≥5% blasts in the bone marrow and/or persistence or reappearance of peripheral blasts. Patients who, upon central review, have <5% blasts in the bone marrow at baseline may be replaced to ensure enough patients for the efficacy analyses.

   In addition, all patients must have:
4. White blood cell (WBC) count below 25,000/μL at time of enrolment. Patients may receive cytoreduction prior to enrolment per Inclusion Criteria 12 and 15
5. Male or female patients aged ≥18 years of age
6. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2
7. Adequate cardiac function defined as ejection fraction (EF) of ≥45% by echocardiogram or multigated acquisition (MUGA) scan.

   Prior Therapy:
8. Prior treatment-related toxicities must have resolved to ≤Grade 1 before enrolment, except for ≤Grade 2 neuropathy or alopecia.
9. Radiation therapy: ≥60 days since TBI, craniospinal, or ≥50% pelvic radiation; ≥14 days since local palliative (small port) radiation.
10. Stem cell infusion: ≥90 days since HSCT and ≥4 weeks since DLI.
11. Immunotherapy: ≥28 days since prior immunotherapy (including tumor vaccines) and ≥21 days since CAR T-cell or other modified T/NK cell therapy.
12. Antileukemia therapy: ≥14 days or 5 half-lives (whichever is shorter) since last antileukemia therapy (e.g. small molecule, cytotoxic, or myelosuppressive therapy), unless otherwise specified. Hydroxyurea for cytoreduction can be initiated without restriction related to timing of study entry. Hydroxyurea can be continued concomitantly with GB3226. Please also refer to Appendix 6 that includes treatment options for the treatment of Differentiation Syndrome.

    Patients may receive intrathecal chemotherapy at the time of diagnostic lumbar puncture at least 24 hours prior to the start of GB3226 and may continue prophylactic intrathecal chemotherapy beginning in Cycle 2 at the treating physician's discretion.
13. Hematopoietic growth factors: ≥7 days since short-acting and ≥14 days since long-acting growth factor therapy.
14. Biologics: ≥90 days or 5 half-lives (whichever is shorter) since antineoplastic biologic therapy.
15. Steroids: ≥7 days since systemic glucocorticoids, except for physiologic doses (≤10 mg prednisone daily) or if used as cytoreductive therapy.
16. Adequate liver and kidney function i.e., i) Estimated glomerular filtration rate (GFR) based on local institutional practice (e.g., Cockcroft-Gault formula) ≥ 60 mL/min/1.73m2 ii) Adequate liver function defined as: Total bilirubin <1.5 times the upper limit of normal (ULN) or normal conjugated bilirubin, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 times ULN (unless attributed to leukemic involvement).

    Contraception
17. Female of childbearing potential: willing to use a highly effective method of contraception or double barrier method from the time of enrolment through 180 days following the last study drug dose.
18. childbearing potential males with female partners of agrees to use barrier contraception from the time of enrolment through 90 days following the last study drug dose.

    Informed Consent
19. Patient is able and willing to provide written informed consent and able to follow study instructions.

Exclusion Criteria

Patients meeting any of the following criteria are NOT eligible for study participation:

Diagnosis

1. Diagnosis of active acute promyelocytic leukemia. (APML)
2. Diagnosis of chronic myelogenous leukemia (CML) in blast crisis
3. Active CNS disease (cytology, such as any blasts on cytospin, or radiography). Patients who have cleared CNS disease by at least one negative tap prior to dosing may be enrolled, and prophylactic intrathecal chemotherapy may be continued while on trial.

   The following patients are required to have a lumbar puncture or Ommaya reservoir tap during the screening period:
   1. Signs and symptoms of CNS disease
   2. AML with monocytic phenotype
   3. WBC ≥50,000 μL at disease presentation
   4. History of CNS or any extramedullary disease Infection
4. Detectable human immunodeficiency virus (HIV) viral load within the previous 6 months. Patients with a known history of HIV 1/2 antibodies must have viral load testing prior to study enrolment.
5. Hepatitis B (defined as hepatitis B virus [HBV] surface antigen positive and HBV core antibody positive, or positive HBV deoxyribonucleic acid [DNA]).
6. Hepatitis C (defined as positive hepatitis C [HCV] antibody with reflex to positive HCV ribonucleic acid [RNA]).

   NB: Patients with controlled HIV, Hep B and Hep C disease will not be excluded from study enrolment.

   Pregnancy and Breast-Feeding
7. Pregnant or nursing women. Negative serum pregnancy tests are required during Screening and a negative serum or urine pregnancy test is required within 72 hours prior to receiving the first study drug administration, in females of childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Concurrent Conditions

   Cardiac Disease:
8. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥III), life-threatening, uncontrolled hypertension or arrhythmia, ischemic or severe valvular heart disease, cerebrovascular accident, or transient ischemic attack.
9. Mean QTcF ≥450 ms for males or ≥470 ms for females on triplicate ECG. Appropriate corrections for patients with bundle branch block and those on pacemakers are allowed.

   Gastrointestinal Disease:
10. Any gastrointestinal issue of the upper GI tract likely to affect oral drug absorption or ingestion (e.g., gastric bypass, gastroparesis, etc.).
11. Cirrhosis with a Child-Pugh score of B or C.
12. Graft-Versus-Host Disease (GVHD): Signs or symptoms of acute or chronic GVHD > Grade 2 within 4 weeks of enrolment. All transplant patients must have been off all systemic immunosuppressive therapy and calcineurin inhibitors for at least 4 weeks prior to enrolment. Patients may be on physiological doses of steroids (≤10 mg/day).
13. Concurrent malignancy in the previous 2 years, with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ, melanoma in situ) treated with potentially curative therapy, or concurrent low-grade lymphoma, that is asymptomatic and lacks bulky disease and shows no evidence of progression, and for which the patient is not receiving any systemic therapy or radiation.
14. Concurrent malignancy must be in complete remission (CR) or no evidence of disease (NED) during this timeframe.
15. Pre-existing disorder predisposing the patient to a serious or life-threatening infection (e.g. cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias not related to AML).
16. Acute or chronic systemic fungal, bacterial, viral, or other infection which is uncontrolled.
17. Major surgery within 4 weeks prior to the first dose of GB3226.
18. History of or any concurrent condition, therapy, laboratory abnormality, or allergy to excipients (see formulation details in Investigator Brochure) that in the Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.

    Concomitant Medications and Interventions
19. Any commercially available or investigational antileukemic therapy other than GB3226, with the following exceptions:

    * Short-term administration of corticosteroids and/or hydroxyurea for cytoreduction. Alternative cytoreductive agents as judged by the treating physician after consultation with study physician may be applied - see also Appendix 6.
    * Intrathecal chemotherapy for CNS prophylaxis is permitted, at the treating physician's discretion. In the Phase 1 DLT evaluable cohort, CNS prophylaxis may continue starting in C2D1.
    * Receipt of an investigational agent within 30 days of starting GB3226, unless inclusion criteria 9-13, then the longer period must be applied. Patients may continue with noninterventional follow-up from previous clinical studies.
    * Any concurrent systemic treatment to prevent GVHD.
20. The following Exclusions apply related to concomitant use of CYP3A4 inhibitors or inducers:

Phase 1:

Cohort A: Arm E: Concurrent use of weak, moderate, and strong inhibitors or inducers of CYP3A4, which should be discontinued at least 7 days prior to enrolment.

Cohort B: Concurrent use of weak, moderate and strong CYP3A4 inhibitors/inducers (except for systemic itraconazole, ketoconazole, posaconazole, or voriconazole, which should have been started at least 7 days prior to enrolment). Other weak, moderate or strong inhibitors or inducers of CYP3A4 should be discontinued at least 7 days prior to enrolment Cohort C: Concurrent use of weak, moderate, and strong inhibitors or inducers of CYP3A4, except for isovuconazole or fluconazole, which should have been started at least 7 days prior to enrolment. All other CYP3A4 inhibitors should be discontinued at least 7 days prior to enrolment.

Phase 2:

Patients who will not be receiving GB3226 in combination with a CYP3A4 inhibitor antifungal must discontinue all CYP3A4 inhibitors at least 7 days prior to the first dose of GB3226. These patients will receive the GB3226 RP2D established for administration without a CYP3A4 inhibitor as determined in the Phase 1 part of the study.

Patients who will be receiving GB3226 in combination with a CYP3A4 inhibitor antifungal must have initiated the antifungal treatment at least 24 hours prior to enrolment. These patients will receive the GB3226 RP2D established for co-administration with a CYP3A4 inhibitor as determined in the Phase 1 part of the study.

Note: The RP2D for GB3226 for patients on a CYP3A4 inhibitor versus patients who are not on a CYP3A4 inhibitor may be different.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-06-10 (Estimated); Primary Completion 2029-06-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (Phase 1) | 28 Days
  Incidence of dose-limiting toxicities events identified
To assess the safety and tolerability of GB3226 | 28 Days
  Incidence of adverse events as reported by investigators.
To characterize the PK parameters of GB3226 | 28 Days
  Plasma concentrations of GB3226
To assess the complete remission and complete remission with partial hematologic recovery rate (Phase 2) | 28 Days
  Number of subjects in complete remission or complete remission with partial hematologic recovery